CLINICAL TRIAL: NCT01697995
Title: Diagnostic and Prognostic Value of the Stress Induced Right Ventricular Uptake on Lexiscan Stress MPI in Patients With Known or Suspected Coronary Artery Disease (CAD).
Brief Title: Stress Induced Right Ventricular Uptake on Lexiscan Stress MPI
Acronym: RVuptakeLexi
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Aiden Abidov (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor-Investigator, Aiden Abidov, Associate Professor of Medicine and Radiology, University of Arizona
Organization: University of Arizona (Other)
Other Study IDs: REGA-11J08
Record Dates: First submitted 2012-08-06; First posted 2012-10-02 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Increased Right Ventricular Radiotracer Uptake
Keywords: right ventricle; radiotracer uptake; Myocardial Perfusion Imaging; balanced ischemia

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lexiscan-Echo echo subjects: No Intervention: Observational study
- Lexiscan-Echo control subjects: No intervention: observational study

SUMMARY:
The objectives of this study are to determine the:

1. Diagnostic value of stress induced RV changes on Lexiscan stress MPI as compared to Exercise stress MPI in predicting a significant CAD.
2. Prognostic value of stress induced RV changes on Lexiscan stress MPI in predicting adverse short-term and long-term clinical outcomes after the index test.

DETAILED DESCRIPTION:
Phase 1: Retrospective data collection/analysis All Lexiscan and exercise MPI images on patients performed for clinical indications in calendar year 2010 who had subsequent coronary angiogram within 3 months after index MPI will be retrieved for review by two experts. We will identify different types of RV uptake and RV overload during stress as well as presence or absence of these changes on resting images. Analysis will include increased RV uptake, enlargement, hypertrophy, thinning of RV and flattening of the interventricular septum. Diagnostic performance (sensitivity, specificity and diagnostic accuracy) of the identified pathological RV phenotypes in identifying severe and extensive disease will be evaluated by comparison with contrary angiograms. Comparison of the set of parameters identifying pathological RV changes, identifying normal and abnormal values of these novel ancillary markers, as well as assessing their diagnostic accuracy in patients with suspected and known CAD during vasodilator stress versus exercise stress MPI will be done.

Phase 2: Prospective data validation Patients referred for the Lexiscan stress MPI will be followed prospectively after obtaining an informed consent. All comers after June 1 2012 will be included. Prediction of coronary artery disease will be performed by applying the previously derived pathological RV criteria on the prospective stress MPIs. 2D-Echocardiogram will be performed for all the patients who do not have an Echocardiogram performed for clinical indication within 1 month of their index Lexiscan stress MPI. We will also include 100 patients referred for the exercise stress MPI who will serve as controls.

All patients will be prospectively followed up for a total of 12 months for the following prognostic end points:

1. Hard cardiac events (cardiac death or MI);
2. Total (all-cause) mortality;
3. Cardiovascular hospitalization rate. Cardiac death (CD) will be defined as death attributable to any cardiac cause (eg, lethal arrhythmia, myocardial infarction [MI], or pump failure) as confirmed by review of death certificate and medical records.

ELIGIBILITY:
Inclusion Criteria:

1. Retrospective population (approximately 300 charts to be reviewed)

   * Patients with MPI and 2D Echocardiogram within one month of the stress testing in calendar year 2010 at University Medical Center, Tucson AZ.
   * 18 years or older.
2. Prospective population (approximately 350 subjects to be recruited)

   * Patients scheduled for MPI at University Medical Center, Tucson AZ.
   * 18 years to 89 years old

Exclusion Criteria (applied to both retrospective and prospective arms):

* patients with nondiagnostic or technically defective MPI
* incomplete clinical data
* severe valvular heart disease
* complex congenital heart disease
* life expectancy less than one year at the time of the index MPI
* unable to follow up (absence of permanent address)
* Known prisoners, pregnant women and cognitively impaired patients.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Retrospective population (approximately 300 charts to be reviewed)
     * Patients with MPI and 2D Echocardiogram within one month of the stress testing in calendar year 2010 at University Medical Center, Tucson AZ.
     * 18 years or older
  2. Prospective population (approximately 350 subjects to be recruited)
     * Patients scheduled for MPI at University Medical Center, Tucson AZ, and invited to participate in this study.
     * 18 years to 89 years old
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Hard cardiac events (cardiac death or MI) | within 1 year after the index test
  Patient follow-up evaluated for hard cardiac events (cardiac death or MI)in the year post index test determined by telephone interviews or review of medical records

SECONDARY OUTCOMES:
Total (all-cause) mortality | within 1 year after the index test
  Total (all-cause) mortality in the year post index test determined by telephone interviews or review of medical records
Cardiovascular hospitalization rate | within 1 year after the index test
  Cardiovascular hospitalization rate in the year post index test determined by telephone interviews or review of medical records

CONTACTS AND LOCATIONS:
Overall Officials: Aiden Abidov, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Medical Center, Tucson, Arizona, United States